CLINICAL TRIAL: NCT06813352
Title: Analysis of Facial Expressions for Pain Recognition: Using Artificial Intelligence and Biomarkers as a Pain Diagnostic Tool in Fibromyalgia, a Pilot Study
Brief Title: Analysis of Facial Expressions for Pain Recognition in Fibromyalgia: Using Artificial Intelligence and Biomarkers
Acronym: Fibromyalgia
Status: Recruiting | Type: Observational
Sponsor: Faculdade de Ciências Médicas de Minas Gerais (Other)
Collaborators: Fundação de Amparo à Pesquisa do estado de Minas Gerais (Other); Conselho Nacional de Desenvolvimento Científico e Tecnológico (Other Government)
Responsible Party: Principal Investigator, Alessandra Hubner de Souza, Main supervisor of the study, statistical analyst and specialist in pain studies; pHd IN Pharmacological Sciences, Faculdade de Ciências Médicas de Minas Gerais
Other Study IDs: CMMG
Record Dates: First submitted 2024-12-19; First posted 2025-02-06 (Actual); Last update posted 2025-11-19 (Actual); Status verified 2025-02

CONDITIONS: Fibromyalgia (FM); Pain; Catastrophizing Pain
Keywords: Fibromyalgia; Artificial intelligence; Molecular biomarkers; Catastrophism; Facial expression
MeSH Terms: conditions — Fibromyalgia; Pain; Facial Expression

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Patient Registry: Yes
Target Follow-Up Duration: 1 Day
Biospecimen Retention: Samples With DNA — Biological samples of saliva.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Patients diagnosed with fibromyalgia: The aim is to follow fibromyalgia patients over a period of months to analyze pain intensity and identify molecular markers associated with the condition. The study encompasses facial analysis techniques and molecular markers, along with artificial intelligence tools, to quantify pain and understand the underlying mechanisms of fibromyalgia. The methodology is predominantly quantitative, focused on collecting and analyzing objective data on pain and associated markers.
- Patients without a diagnosis of fibromyalgia: The aim is to follow patients with pain over a period of months to analyze the intensity and identify molecular markers associated with the condition. The study encompasses facial analysis techniques and molecular markers, along with artificial intelligence tools, to quantify pain and understand the underlying mechanisms of fibromyalgia. The methodology is predominantly quantitative, focused on collecting and analyzing objective data on pain and associated markers.

SUMMARY:
Fibromyalgia (FM) is a chronic musculoskeletal pain syndrome with characteristics of generalized body pain, low pain threshold, tenderness and stiffness in muscles, tendons and joints. The assessment of pain in this condition is a challenge due to its subjective nature. A promising approach to assessing pain intensity is facial expression analysis, which can serve as an objective indicator. In addition, research seeks to identify molecular molecular markers to quantify pain. However, the lack of a standardized system has made it difficult to identify reliable markers. In summary, the search for objective methods of assessing pain in fibromyalgia is essential in order to develop more effective more effective treatments. Facial expression analysis and the investigation of molecular markers are promising ways of quantifying pain intensity more accurately and intensity of pain more accurately and reliably in fibromyalgia.

DETAILED DESCRIPTION:
Introduction:

Fibromyalgia (FM) is a chronic syndrome characterized by diffuse musculoskeletal pain, fatigue and sleep disturbances, with a major impact on quality of life. Due to the subjectivity of pain assessment, the development of objective methods is essential. This study explores the use of artificial intelligence (AI) in the analysis of facial expressions, combined with the investigation of molecular markers, as an innovative and quantitative approach to pain assessment in patients with FM.

Objective:

To validate the application of an AI tool combined with facial expression analysis and molecular biomarker research to measure pain intensity in FM patients.

Methodology:

An observational cohort study was carried out with 122 participants, divided into two groups: patients with FM (n=61) and without FM (n=61). Data collection included:

1. Facial expression recording: A convolutional neural network algorithm was used to analyze facial patterns associated with pain.
2. Biological samples: 1mL of saliva will be collected from each participant using the salivette method and processed to extract DNA, RNA and plasma proteins. The proteins will be quantified by ELISA and the genes associated with FM will be analyzed by RT-qPCR.
3. Clinical Questionnaires: Psychometric instruments such as the Visual Analogue Scale (VAS) and the Generalized Pain Index (GDI) were used to validate the results.
4. Statistical analysis: The data was analyzed using Kappa and Bland-Altman correlations to assess the agreement between the AI methods and the questionnaires, with a significance level of p<0.05.

The AI algorithm will use consistent facial patterns correlating them to the reported pain intensity, in agreement (Kappa=0.82) with the results of the clinical scales.The molecular markers analyzed are expected to show significant differences between the groups, with increased expression of inflammatory proteins in FM patients (p<0.05). The integration of facial and molecular analysis aims to amplify the accuracy of pain intensity classification.

This approach represents a promising advance in the diagnosis and management of the syndrome, contributing to personalized therapies and improving patients' quality of life.

ELIGIBILITY:
Inclusion Criteria:

* The inclusion criteria are patients with no diagnosed cognitive deficit and who are willing to take part in the study.

Exclusion Criteria:

* Exclusion criteria are patients who use medication that can affect anxiety or depression or inability to understand the instructions.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: The study will be carried out with adult patients aged between 18 and 65 diagnosed with fibromyalgia at the outpatient clinic of the Faculdade Ciências Médicas de Minas Gerais and Clínica Ampla de Reumatologia in Belo Horizonte. The inclusion criteria were patients with no diagnosed cognitive deficit and who were willing to take part in the study. The exclusion criteria are patients who use medication that can affect anxiety or depression or who are unable to understand the instructions. Thus, once the patients agree to participate, they will be asked to sign the Informed Consent Form (ICF), which will provide detailed information about the nature of the study, the criteria for participation, the possible risks and benefits involved.
Sampling Method: Probability Sample
Enrollment: 122 (Estimated)
Dates: Start 2025-11-17 (Actual); Primary Completion 2026-02-01 (Estimated); Study Completion 2026-09-01 (Estimated)

PRIMARY OUTCOMES:
Use the artificial intelligence tool to analyze the facial expression of patients with fibromyalgia in order to recognize pain. | The estimated time for the anamnesis is one hour, during which time biological samples will be taken and each patient's facial expressions will be recorded on camera.
  Use the artificial intelligence tool to analyze the facial expression of patients with fibromyalgia in order to recognize pain. 61 patients with fibromyalgia will be compared with 61 patients without fibromyalgia.

SECONDARY OUTCOMES:
Biochemical analysis of biomarkers in the detection of pain in fibromyalgia. | Estimated collection and analysis time: 5 hours of durability
  122 samples containing 1ml of saliva will be collected in order to check for changes in oxidative stress and nociceptive markers (by spectrophotometry and ELISA).

CONTACTS AND LOCATIONS:
Locations (1):
- Outpatient Faculty Medical Sciences, Belo Horizonte, Minas Gerais, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Barua VB, Juel MAI, Blackwood AD, Clerkin T, Ciesielski M, Sorinolu AJ, Holcomb DA, Young I, Kimble G, Sypolt S, Engel LS, Noble RT, Munir M. Tracking the temporal variation of COVID-19 surges through wastewater-based epidemiology during the peak of the pandemic: A six-month long study in Charlotte, North Carolina. Sci Total Environ. 2022 Mar 25;814:152503. doi: 10.1016/j.scitotenv.2021.152503. Epub 2021 Dec 23. PMID 34954186
- [Background] Agarwal A, Emary PC, Gallo L, Oparin Y, Shin SH, Fitzcharles MA, Adachi JD, Cooper MD, Craigie S, Rai A, Wang L, Couban RJ, Busse JW. Physicians' knowledge, attitudes, and practices regarding fibromyalgia: A systematic review and meta-analysis of cross-sectional studies. Medicine (Baltimore). 2024 Aug 2;103(31):e39109. doi: 10.1097/MD.0000000000039109. PMID 39093781
- [Background] Ahmad M, Ahmed I, Jeon G. A sustainable advanced artificial intelligence-based framework for analysis of COVID-19 spread. Environ Dev Sustain. 2022 Aug 16:1-16. doi: 10.1007/s10668-022-02584-0. Online ahead of print. PMID 35993085